CLINICAL TRIAL: NCT02904356
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Obsessive-Compulsive Disorder (OCD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAQ8771
Record Dates: First submitted 2016-08-25; First posted 2016-09-19 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; TMS; Neuromodulation; Obsessive-Compulsive Disorder; Transcranial Magnetic Stimulation; Imaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Brainsway H-coil for rTMS (Experimental): Brainsway H-coil for repetitive transcranial magnetic stimulation: High-frequency rTMS will be administered to the medial prefrontal cortex for 3 weeks.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — High-frequency, brainsway H-coil for repetitive transcranial magnetic stimulation will be administered to the medial prefrontal cortex for 3 weeks. The intensity of stimulation will be based on resting-motor threshold (RMT).
  Other Names: rTMS

SUMMARY:
The study aims to assess the impact of repetitive transcranial magnetic stimulation (rTMS) on brain imaging and neurophysiological measures of cognitive control in patients with Obsessive-Compulsive Disorder (OCD).

DETAILED DESCRIPTION:
With a prevalence of nearly 3%, obsessive-compulsive disorder (OCD) is one of the most common psychiatric disorders in the US. The first line of treatment for OCD comprises pharmacotherapy with serotonin reuptake inhibitors (SRIs) and cognitive behavioral therapy (CBT). Although adherence to these therapies has been shown to improve symptoms in at least half of patients, some have residual symptoms and a small percentage are refractory to standard therapies. Transcranial magnetic stimulation (TMS) may offer an alternate, less-invasive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Obsessive Compulsive Disorder, as confirmed by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) (SCID).
* Subjects should have at least a moderate level of OCD severity as defined by a Yale-Brown Obsessive Compulsive Disorder Scale (YBOCS) score of ≥ 20.

Exclusion Criteria:

* Individuals diagnosed by the investigators with the following conditions: Bipolar Disorder (lifetime), any Psychotic Disorder (lifetime), history of substance abuse or dependence within the past year (expect nicotine and caffeine).
* An Axis II Personality Disorder, which in the judgment of the investigator may hinder the patient in completing the procedures required by the study protocol.
* Individuals with a clinically defined neurological disorder including, but not limited to: stroke, tics, space occupying brain lesion, any history of seizures except those therapeutically induced by electroconvulsive therapy (ECT), history of cerebrovascular accident, transient ischemic attack within two years, cerebral aneurysm, dementia, Parkinson's Disease, Huntington Chorea, Multiple Sclerosis.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for >5 minutes.
* History of treatment with rTMS therapy for any disorder.
* History of treatment with Deep Brain Stimulation.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* Current illicit drug use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Sheth, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brainsway H-coil for rTMS
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brainsway H-coil for rTMS
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
Diagnosis of Obsessive Compulsive Disorder [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Magnetic Resonance Imaging (fMRI) BOLD Response
Description: Change in blood-oxygen-level dependent (BOLD) correlates corresponding to task engagement before and after rTMS will be assessed.
Time Frame: Up to 1 month
Population: PI left institution, no data was collected and analyzed in the specified manner.
Arm/Group | Brainsway H-coil for rTMS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 month.
Arm/Group | Brainsway H-coil for rTMS
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
PI left institution, no data was collected and analyzed in the specified manner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT02904356/Prot_SAP_000.pdf